CLINICAL TRIAL: NCT03911752
Title: Approach to Sexuality From Occupational Therapy in People With Acquired Bran Injury in Subacute Stage
Brief Title: Approach to Sexuality From Occupational Therapy in People With Acquired Brain Injury in Subacute Stage
Status: Completed | Type: Observational
Sponsor: Universidade da Coruña (Other)
Collaborators: University Hospital A Coruña (Other)
Responsible Party: Principal Investigator, Thais Pousada, PhD Health Science. Occupational Therapist, Universidade da Coruña
Other Study IDs: 2017/587
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Results first posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-10

CONDITIONS: Occupational Therapy; Sexuality; Acquired Brain Injury
Keywords: Occupational Therapy; Sexuality; Acquired Bain Injury; Subacute Stage; Qualitative Study
MeSH Terms: conditions — Sexuality; Brain Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- People with Acquired Brain Injury: People with Acquired Brain Injury in a subacute stage who go to occupational therapy (N=8).
  Interventions: Other: Semi-structured interviews; Other: Canadian Occupational Performance Measure
- Partners of people with Acquired Brain Injury: Partners of people with Acquired Brain Injury in a subacute stage who go to occupational therapy (N=2).
  Interventions: Other: Semi-structured interviews
- Relatives of people with Acquired Brain Injury: Relatives of people with Acquired Brain Injury in a subacute stage who go to occupational therapy (N=2).
  Interventions: Other: Semi-structured interviews

INTERVENTIONS:
Other: Semi-structured interviews — Semi-structured interviews were used to obtain the main data in this study.
Other: Canadian Occupational Performance Measure — The Canadian Occupational Performance Measure was used with the group of people with Acquired Brain Injury to know their occupational priorities.
  Other Names: COPM
  Groups: People with Acquired Brain Injury

SUMMARY:
Objectives: To analyse if people with acquired brain injury in sub-acute situation, as well as their relatives, and/or partners, consider relevant the approach to sexuality during their Occupational Therapy intervention.

Methodology: This study presents a qualitative design with a phenomenological approach. Twelve participants were interviewed: eight people with acquired brain injury, two relatives and two partners who agreed to participate. The information has been collected through interviews.

ELIGIBILITY:
People with Acquired Brain Injury

Inclusion Criteria:

* Being over 18 years.
* Have a diagnosis framed within the concept of Acquired Brain Injury.
* To be in the sub-acute stage after the Acquired Brain Injury.
* Take Occupational Therapy to the Neurology Service of the Rehabilitation Unit of the Maritime Hospital of Oza (CHUAC) for a minimum of two months.

Exclusion Criteria:

* Do not accept to participate in the study.
* Present a decrease in the level of consciousness.
* Present alterations at the cognitive level that suppose a score of less than 20 on the Mini-mental State Examination (MMSE).
* Present disinhibition after acquired brain damage.
* Present sensory aphasia.

Partners and relatives of people with Acquired Brain Injury

Inclusion Criteria:

* Being over 18 years.
* Being partner or relative of a person who has a diagnosis framed within the concept of Acquired Brain Injury.
* Being partner or relative of a person who is in the sub-acute stage after the Acquired Brain Injury.
* Being partner or relative of a person who takes Occupational Therapy to the Neurology Service of the Rehabilitation Unit of the Maritime Hospital of Oza (CHUAC) for a minimum of two months.

Exclusion Criteria:

* Do not accept to participate in the study.
* Present a decrease in the level of consciousness.
* Present alterations at the cognitive level that suppose a score of less than 20 on the Mini-mental State Examination (MMSE).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who go to Maritime Hospital of Oza (University Hospital Complex of A Coruña) because it is a person with Acquired Brain Injury or a relative or partner of a person with these characteristics
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thais Pousada García, Principal Investigator — PhD Health Science. Occupational Therapist.
Locations (1):
- Faculty of Health Sciences. University of A Coruña, A Coruña, Galicia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haag HL, Caringal M, Sokoloff S, Kontos P, Yoshida K, Colantonio A. Being a Woman With Acquired Brain Injury: Challenges and Implications for Practice. Arch Phys Med Rehabil. 2016 Feb;97(2 Suppl):S64-70. doi: 10.1016/j.apmr.2014.12.018. Epub 2015 Feb 7. PMID 25666783
- [Background] Schmitz MA, Finkelstein M. Perspectives on poststroke sexual issues and rehabilitation needs. Top Stroke Rehabil. 2010 May-Jun;17(3):204-13. doi: 10.1310/tsr1703-204. PMID 20797965
- [Background] Moreno JA, Arango Lasprilla JC, Gan C, McKerral M. Sexuality after traumatic brain injury: a critical review. NeuroRehabilitation. 2013;32(1):69-85. doi: 10.3233/NRE-130824. PMID 23422460
- [Background] Brunsden C, Kiemle G, Mullin S. Male partner experiences of females with an acquired brain injury: An interpretative phenomenological analysis. Neuropsychol Rehabil. 2017 Sep;27(6):937-958. doi: 10.1080/09602011.2015.1109525. Epub 2015 Nov 26. PMID 26610187
- [Background] Townsend E, Wilcock AA. Occupational justice and client-centred practice: a dialogue in progress. Can J Occup Ther. 2004 Apr;71(2):75-87. doi: 10.1177/000841740407100203. PMID 15152723
- [Background] McGrath M, Lynch E. Occupational therapists' perspectives on addressing sexual concerns of older adults in the context of rehabilitation. Disabil Rehabil. 2014;36(8):651-7. doi: 10.3109/09638288.2013.805823. Epub 2013 Jun 26. PMID 23802139
- [Background] Hyland A, Mc Grath M. Sexuality and occupational therapy in Ireland--a case of ambivalence? Disabil Rehabil. 2013 Jan;35(1):73-80. doi: 10.3109/09638288.2012.688920. Epub 2012 Jun 2. PMID 22657159
- See also: World Health Organization (WHO). Defining sexual health [Internet]. WHO. World Health Organization; 2018 — http://www.who.int/reproductivehealth/topics/sexual_health/sh_definitions/en/
- See also: Sakellariou D, Simó Algado S. Sexuality and Disability: a Case of Occupational Injustice. Br J Occup Ther. 2006;69(2):69-76. — https://www.researchgate.net/publication/227944687_Pollard_N_Sakellariou_D_2007_Sex_and_occupational_therapy_contradictions_or_contraindications_British_Journal_of_Occupational_Therapy_70_8_361-5
- See also: Ministerio de Sanidad, Política Social e Igualdad. Estrategia Nacional de Salud Sexual y Reproductiva. [Internet]. 2011. p. 178. — http://www.msc.es/organizacion/sns/planCalidadSNS/pdf/equidad/ENSSR.pdf
- See also: Jones B. S, Duarte B. T, Astorga U. N, Pardo M, Sepúlveda R. Aproximación a la experiencia de cuerpo y sexualidad de un grupo de mujeres chilenas con discapacidad física congénita. Rev chil ter ocup. 2015;15(1):19-32. — http://repositorio.uchile.cl/bitstream/handle/2250/151907/24-Aproximacion-a-la-experiencia-de-cuerpo-y-sexualidad.pdf?sequence=1&isAllowed=y
- See also: Federación Española de Daño Cerebral. Talleres y Cuadernos FEDACE sobre Daño Cerebral Adquirido. 1.a ed. de la Cruz Martín-Romo C, Rubio Arribas N, editores. Madrid: FEDACE; 2010. 1-170 p. — http://sexualidadydiscapacidad.es/wp-content/uploads/Sexualidad-y-Da%C3%B1o-Cerebral-Adquirido_DCA_-Cuadernos-FEDACE_Natalia-Rubio-y-Carlos-de-la-Cruz_2010.pdf
- See also: Cortes Generales del Reino de España. Ley Orgánica 2/2010, de 3 de marzo, de salud sexual y reproductiva y de la interrupción voluntaria del embarazo. Boletín Of del Estado. 2010;55(3514):21001-14. — https://www.boe.es/buscar/pdf/2010/BOE-A-2010-3514-consolidado.pdf
- See also: Pollard N, Sakellariou D. Sex and Occupational Therapy: Contradictions or Contraindications ? Br J Occup Ther. 2007;70(June 2016):361-5. — https://www.academia.edu/7551382/Sex_and_occupational_therapy_contradictions_or_contraindications
- See also: Moruno P, Agudo P. Análisis teórico de los conceptos privación, alienación y justicia ocupacional. Rev Ter Ocup Galicia [Internet]. 2012;9:44-68. — http://www.revistatog.com/mono/num5/teorico.pdf
- See also: Asociación Española de Medicamentos y Productos Sanitarios. Normas de buena práctica clínica. Guía de buena práctica clínica España; 2002 p. 1-57. — https://www.aemps.gob.es/industria/inspeccionBPC/docs/guia-BPC_octubre-2008.pdf
- See also: Jefatura del Estado. Ley Orgánica 15/1999, de 13 de diciembre, de Protección de Datos de Carácter Personal. BOE España; 1999 p. 43088-99. — https://www.boe.es/buscar/doc.php?id=BOE-A-1999-23750
- See also: Ministerio de Educación, Cultura y Deporte. Orden SSI/81/2017, de 19 de enero, por la que se publica el Acuerdo de la Comisión de Recursos Humanos del Sistema Nacional de Salud. España: Boletín Oficial Del Estado; 2017. — https://www.boe.es/diario_boe/txt.php?id=BOE-A-2017-1200
- See also: Salgado A.C. Investigación cualitativa: diseños, evaluación del rigor metodológico y retos. Liberabit. 2007;13(2006):3-10. — http://www.scielo.org.pe/scielo.php?script=sci_arttext&pid=S1729-48272007000100009
- See also: Sáez S. El hombre "en" la discapacidad física. En: Martínez Sola F, editor. La erótica del encuentro. 1.a ed. Gijón, Spain: COCEMFE ASTURIAS; 2003. p. 33-48. — https://www.cocemfeasturias.es/archivos/251_discapacidad-vida-sexual--la-erotica-encuentro-.pdf
- See also: Cantero Garlito PA, Emeric Méaulle D, Zango Martín I, Domínguez Vega E. Ocupaciones de Mujer(es), ocupaciones de hombre(s): la influencia del sexo sobre la ocupación y sobre la profesión de la terapia ocupacional en España. Rev TOG. 2012;9:96-124. — http://www.revistatog.com/mono/num5/genero.pdf
- See also: Sociedad Española de Geriatría y Gerontología. El 89% de los cuidadores en España son mujeres y en el 47% de los casos, el cuidador principal es un familiar. [Internet]. Sociedad Española de Geriatría y Gerontología. 2016. p. 1 — https://www.segg.es/institucional/2016/11/03/el-89-por-ciento-de-los-cuidadores-en-espa%C3%B1a-son-mujeres-y-en-el-47-por-ciento-de-los-casos-el-cuidador-principal-es-un-familiar
- See also: Pizarro Pedraza A. Tabú y eufemismo en la ciudad de Madrid. Estudio sociolíngüístico-cognitivo de los conceptos sexuales. Universidad Complutense de Madrid; 2014. — https://eprints.ucm.es/24937/1/T35255.pdf
- See also: Varela Salgado M, Paz Esqueje J. Resultados de una encuesta sobre educación sexual y hábitos sexuales de los gallegos. Rev Int Androl. 2007;5(2):161-6. — https://www.researchgate.net/publication/250778837_Resultados_de_una_encuesta_sobre_educacion_sexual_y_habitos_sexuales_de_los_gallegos
- See also: Shildrick M. Contested pleasures: The sociopolitical economy of disability and sexuality. Sex Res Soc Policy. 2007;4(1):53-66. — https://www.researchgate.net/publication/225324290_Contested_pleasures_The_sociopolitical_economy_of_disability_and_sexuality

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | People With Acquired Brain Injury | Partners of People With Acquired Brain Injury | Relatives of People With Acquired Brain Injury
Started | 8 | 2 | 2
Completed | 8 | 2 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | People With Acquired Brain Injury | Partners of People With Acquired Brain Injury | Relatives of People With Acquired Brain Injury | Total
Number analyzed (Participants) | 8 | 2 | 2 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 2 | 2 | 12
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 6
  Male | 5 | 0 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 2 | 2 | 12
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 8 | 2 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Felt The Approach to Sexuality During Occupational Therapy is Relevant
Description: 12 semi-structured interviews Qualitative data analysis - Theoretical concept saturation and thematic analyses.
Time Frame: 2 months
Population: Transcription, listening and categorizing the speaking of participants from their answers to the interviews.
Measure: Count of Participants; unit: Participants
Arm/Group | People With Acquired Brain Injury | Partners of People With Acquired Brain Injury | Relatives of People With Acquired Brain Injury
Number analyzed (Participants) | 8 | 2 | 2
Participants | 8 | 2 | 2

2. Primary Outcome: Number of Participants That Identified Having Occupational Priorities
Description: The semi-structured interview Canadian Measure of Occupational Performance (CMOP) was used.
  The COPM measures performance and satisfaction in self-care, productivity and leisure from the client's perspective Areas of everyday living explored during the interview include self-care, productivity or leisure and the occupational performance problems experienced in everyday living are identified.
  In step two, the client is asked to rate the importance of each of the occupations to his/her life using a 10-point rating scale.
  In the third step, the client chooses up to five of the most important problems identified in step two.
  In step four, the client is asked to use a 10 point scale to rate their own level of performance and satisfaction with performance for each of the five problems. These typically range between 1 and 10, where 1 indicates poor performance and low satisfaction, respectively, while 10 indicates very good performance and high satisfaction.
Time Frame: 2 months
Population: Interviews
Measure: Count of Participants; unit: Participants
Groups:
- Partners of People With Acquired Brain Injury: Partners of people with Acquired Brain Injury in a subacute stage who go to occupational therapy
- Relatives of People With Acquired Brain Injury: Relatives of people with Acquired Brain Injury in a subacute stage who go to occupational therapy
Arm/Group | People With Acquired Brain Injury | Partners of People With Acquired Brain Injury | Relatives of People With Acquired Brain Injury
Number analyzed (Participants) | 8 | 2 | 2
Participants
  Activities of Daily Living | 8 | 2 | 2
  Work and productivity | 5 | 1 | 1
  Leisure | 7 | 2 | 1

3. Primary Outcome: Number of Participants With Problems in Performance in His/Her Daily Life
Description: The semi-structured interview Canadian Measure of Occupational Performance (CMOP) was used.
  The client chooses up to five of the most important problems identified in his/her daily life, and he/she is asked to use a 10 point scale to rate their own level of performance. These typically range between 1 and 10, where 1 indicates poor performance while 10 indicates very good performance.
Time Frame: 2 months
Population: Interviews. Data were not collected for Partners and Relatives because they had not any consequences in their performance due to an Acquired Brain Injury.
Measure: Count of Participants; unit: Participants
Arm/Group | People With Acquired Brain Injury | Partners of People With Acquired Brain Injury | Relatives of People With Acquired Brain Injury
Number analyzed (Participants) | 8 | 0 | 0
Participants
  Activities of Daily Living | 8 |  |
  Work and productivity | 4 |  |
  Leisure | 5 |  |

4. Primary Outcome: Number of Participants Who Are Satisfied With Performance in Areas of Everyday Living.
Description: The semi-structured interview Canadian Measure of Occupational Performance (CMOP) was used.
  The client is asked to use a 10 point scale to rate their own satisfaction during the performance of activities of daily life. Satisfaction refers to the self-perception of the results derived from doing any activity of daily life.
  These typically range between 1 and 10, where 1 indicates low satisfaction, respectively, while 10 indicates high satisfaction.
Time Frame: 2 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | People With Acquired Brain Injury | Partners of People With Acquired Brain Injury | Relatives of People With Acquired Brain Injury
Number analyzed (Participants) | 8 | 0 | 0
Participants
  Activities of Daily Living | 4 |  |
  Work and productivity | 5 |  |
  Leisure | 3 |  |

ADVERSE EVENTS:
Time Frame: Not applicable due to the study design
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored
Arm/Group | People With Acquired Brain Injury | Partners of People With Acquired Brain Injury | Relatives of People With Acquired Brain Injury
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT03911752/Prot_000.pdf